CLINICAL TRIAL: NCT05768490
Title: A Prospective, Multicenter, Randomized, Controlled Clinical Study of Early or Delayed Intervention of Brain Radiotherapy Combined With Almonertinib in EGFR Mutated NSCLC With Brain Metastases
Brief Title: Early or Delayed Intervention of Brain Radiotherapy Combined With Almonertinib in EGFR Mutated NSCLC With Brain Metastases
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Li-kun Chen, Professor of Medicine, Sun Yat-sen University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: B2022-428-01
Record Dates: First submitted 2022-12-12; First posted 2023-03-14 (Actual); Last update posted 2023-03-14 (Actual); Status verified 2023-03

CONDITIONS: Brain Metastases; Radiotherapy; EGFR Activating Mutation
MeSH Terms: conditions — Brain Neoplasms | interventions — aumolertinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- early intervention group of brain radiotherapy (Experimental): the brain radiotherapy started within 1 month of almonertinib the brain radiotherapy here specifically refers to stereotactic radiotherapy
  Interventions: Radiation: brain radiotherapy; Drug: Almonertinib
- late intervention group of brain radiotherapy (Active Comparator): Brain radiotherapy was given within 3 months after brain progression during almonertinib treatment
  Interventions: Drug: Almonertinib

INTERVENTIONS:
Radiation: brain radiotherapy — Patients were randomly divided into two groups, experimental group (early intervention group of brain radiotherapy) : the brain radiotherapy started within 1 month of TKI treatment, the brain radiotherapy here specifically refers to stereotactic radiotherapy; Control group (brain radiotherapy late intervention group) : Brain radiotherapy was given within 3 months after brain progression during TKI treatment.
  Arms: early intervention group of brain radiotherapy
Drug: Almonertinib — almonertinib po 110mg QD

SUMMARY:
This is a prospective, multicenter, randomized, controlled clinical study of NSCLC patients with intracranial oligo-metastatic EGFR-sensitive mutations treated with EGFR-TKI Almonertinib , according to the implementation time of brain radiotherapy. Patients were randomly divided into two groups, experimental group (early intervention group of brain radiotherapy) : the brain radiotherapy started within 1 month of TKI treatment, the brain radiotherapy here specifically refers to stereotactic radiotherapy; Control group (brain radiotherapy late intervention group) : Brain radiotherapy was given within 3 months after brain progression during TKI treatment. The differences in OS,iPFS, PFS, iORR, safety, neurocognitive function and quality of life between the two groups were compared.

ELIGIBILITY:
Inclusion Criteria:

* Patients with histologically or cytologically confirmed non-small cell lung cancer;
* Initial diagnosis of intracranial oligometastases (no treatment after brain metastases) was defined as brain parenchymal metastases confirmed by MRI, the number of intracranial parenchymal metastases was less than 5, and the lesions were 3mm away from the optic nerve and brainstem; There must be at least one measurable lesion with a diameter of 5mm or more in the brain.
* EGFR sensitivity mutation (exon19del or exon21 L858R);
* Anti-EGFR-targeting drugs and other TKI drugs have not been used in the past;
* Age 18-75;

Inclusion criteria:

* A history (past or concurrent) of malignancies in other sites, excluding curable non-melanoma skin cancer and cervical carcinoma in situ;
* The subjects had received brain radiotherapy before enrollment;
* Patients whose lung lesions were surgically evaluated as resectable were not included if there was no metastasis in other parts of the body;
* Received EGFR inhibitors (including small molecule or monoclonal antibody therapy) or systematic anti-tumor therapy before treatment;
* Prior patients with interstitial lung disease, drug-induced interstitial disease, radiation pneumonia requiring hormone therapy, or any clinically proven active interstitial lung disease with idiopathic pulmonary fibrosis found on CT scan at baseline;
* Pregnant and lactating patients;
* MRI contraindicated patients;
* Patients who cannot receive oral administration, need intravenous high-energy nutrition, have undergone previous surgery that interferes with absorption, or have active digestive tract ulcers;
* The researchers judged that brain radiotherapy could not be received because of other head and facial diseases;
* Any unstable systemic disease (including active infection, poorly controlled hypertension, unstable angina, congestive heart failure, liver, kidney or metabolic disease).

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 232 (Estimated)
Dates: Start 2023-03-15 (Estimated); Primary Completion 2028-12-31 (Estimated); Study Completion 2029-12-31 (Estimated)

PRIMARY OUTCOMES:
overall survival | 3 years
  The time from randomization to death from any cause.

SECONDARY OUTCOMES:
intracranial progression free survival | 2 years
  patients were randomized from the time of observation of intracranial disease progression or death from any cause
progression free survival | 2 years
  patients were randomized from the time of observation of systemic disease progression or death from any cause
intracranial objective response rate | 6 months
  proportion of patients with complete or partial response of intracranial lesions

CONTACTS AND LOCATIONS:
Overall Officials: Likun Chen, Principal Investigator — sunyat-sen university cancer center
Locations (1):
- Sun-Yat-Sen university, Guangdong, Guangzhou, China